CLINICAL TRIAL: NCT01863602
Title: Special Drug Use Investigation for LAMICTAL (Long Term)
Brief Title: Special Drug Use Investigation for LAMICTAL® (Long Term)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112728
Record Dates: First submitted 2012-10-04; First posted 2013-05-29 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Subjects prescribed lamotrigine tablets: Subjects with epilepsy with partial seizures, tonic-clonic seizuresm or generalized seizures of Lennox-Gastaut syndrome to whom lamotrigine tablets are administered.
  Interventions: Drug: Lamotrigine tablets

INTERVENTIONS:
Drug: Lamotrigine tablets — Administered for long-term according to the prescribing information in the locally approved label by the authorities.

SUMMARY:
The objectives of this post-marketing surveillance (PMS) are to grasp the actual use of lamotrigine tablets to collect safety information in the long-term use according to seizure type and concomitant antiepileptic drug (AED), and to confirm its efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with epilepsy with partial seizures, tonic-clonic seizuresm or generalized seizures of Lennox-Gastaut syndrome
* Subjects who are treated with lamotrigine tablets

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult (>=15 to <65 years) and pediatric (>=2 to <15 years) subjects with epilepsy with the following seizure type who use lamotrigine tablets
  * Partial seizures
  * Tonic-clonic seizures
  * Generalized seizures of Lennox-Gastaut syndrome
Sampling Method: Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2009-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse drug reactions | 1 year
Occurrence of skin disorder after the start of treatment | 1 year
  Presence or absence of skin disorder and its details after the start of treatment will be investigated as a priority investigation item

SECONDARY OUTCOMES:
Overall improvement of subjects' symptoms | 1 year
  Investigators will assess the overall improvement as "remarkably improved". "improved", "slightly improved", "unchanged" or "worsened" on the basis of the degree of change in frequency of seizures, strength, span and other related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline